CLINICAL TRIAL: NCT03204435
Title: Clinical Trail of Hybrid Operating Technique in Management of Intracranial Aneurysms With Coexistence of Atherosclerotic Intracranial Arterial Stenosis
Brief Title: Hybrid Operating Treatment of Coexistence of Intracranial Aneurysms and Cerebrovascular Stenosis
Acronym: HOT-CIACS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: liuxingju (Other Government)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Sponsor-Investigator, liuxingju, Researcher, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJTTH-005
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Intracranial Aneurysm; Cerebrovascular Stenosis; Atheroscleroses, Cerebral
MeSH Terms: conditions — Intracranial Aneurysm; Intracranial Arteriosclerosis | interventions — Endovascular Procedures; Endarterectomy, Carotid

STUDY DESIGN:
Intervention Model Description: Patients of intracranial aneurysms with coexistence of cerebrovascular stenosis, coincident with inclusion and exclusion criterion, will be distributed into traditional therapy group(control group) and hybrid operating group(test group), and conduct with traditional neurosurgical management or one-stage hybrid operating management separately.
  Traditional therapy group: intervene the aneurysms and vascular stenosis unsimultaneously. Clipping procedure is preferred to aneurysms, while endovascular intervention is preferred to stenosis.
  Hybrid operation group: one-stage hybrid operating technique is conducted. The aneurysms and vascular stenosis will be executed via the cooperation of microsurgical procedure and endovascular interventional techniques.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional therapy (Other): Consists of microsurgical aneurysmal operating techniques, endovascular techniques for intracranial aneurysms, endovascular techniques for cerebrovascular stenosis, and carotid endarterectomy, which are presented by stages.
  Interventions: Procedure: Microsurgical aneurysmal operating techniques; Procedure: endovascular techniques for cerebrovascular stenosis; Procedure: endovascular techniques for intracranial aneurysms; Procedure: carotid endarterectomy
- Hybrid operation (Experimental): Consists of microsurgical aneurysmal operating techniques, endovascular techniques for intracranial aneurysms, endovascular techniques for cerebrovascular stenosis, and carotid endarterectomy, which are presented in one-stage in hybrid operating theater.
  Interventions: Procedure: Microsurgical aneurysmal operating techniques; Procedure: endovascular techniques for cerebrovascular stenosis; Procedure: endovascular techniques for intracranial aneurysms; Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: Microsurgical aneurysmal operating techniques — The microsurgical techniques used to evacuate the aneurysm out of circulation or reduce its risk of rupture by aneurysmal clipping, wrapping,or isolation.
  Other Names: microsurgical aneurysmal clipping; microsurgical aneurysmal wrapping; microsurgical aneurysmal isolation
Procedure: endovascular techniques for cerebrovascular stenosis — The endovascular techniques that recanalize the narrowed or occluded cerebrovascular, including stent implantation, balloon dilatation.
  Other Names: endovascular stenting; endovascular balloon dilatation
Procedure: endovascular techniques for intracranial aneurysms — The endovascular techniques that embolize the cavity of aneurysms to reduce the risk of rupture, including coiling embolization, balloon-assisted occlusion.
  Other Names: endovascular coiling; endovascular balloon occlusion; flow diverter
Procedure: carotid endarterectomy — A microsurgical technique to recanalize the stenosis or occluded proximal segment of carotid artery.

SUMMARY:
To evaluate the clinical benefits and risks of hybrid operating techniques in management of intracranial aneurysms with coexistence of atherosclerotic intracranial arterial stenosis.

DETAILED DESCRIPTION:
Purpose: Have an evaluation of clinical benefits and risks of hybrid operating techniques in management of intracranial aneurysms (IAs) with coexistence of atherosclerotic intracranial arterial stenosis (AIAS), whose management strategies are inconsistent. Meanwhile, as a new cooperative interventional modality, optimized workflows, technical key knots and operation routines will be explored in the study.

Objects: Patients with IAs with coexistence of AIAS, coincident with inclusion and exclusion criterion and admitted in participating organizations.

Methods: Patients will be distributed into 2 groups, including traditional therapy group(control group) and hybrid operating group(trial group), and conduct with traditional multi-stage neurosurgical management or one-stage hybrid operating management correspondingly. The morbidity rate of peri-operative cerebral hemorrhagic/ischemic event is considered to be the primary observing indicator, and morbidity rate of peri-operative cerebral hemorrhagic/ischemic event, while peri-operative mortality rate, and health-economic indicators are secondary indicators.The information of operations will be recorded in detail as evidence of optimization of workflow and technical key knots.

ELIGIBILITY:
Inclusion Criteria:

* For aneurysms:
* with diagnosed complex intracranial aneurysm by digital subtraction angiography(DSA);
* got SAH in history;
* neural functional deficits due to aneurysms;
* with <4 in Hunt-Hess Grades;
* ≥5.0mm in the maximum diameter;
* <70 years old;
* with irregular morphological features and high rupture risk.

and for stenosis

* Intracranial vessels:
* >50% in rate of stenosis with ischemic symptoms/perfusing evidence/lacunar infarction in supplying territory, failed in conservative treatment;
* with a deliverable position of intracranial stents devices.
* or Vertebral arterial system:
* ≥70% in the rate of stenosis, with contralateral vertebral arterial occlusion;
* symptomatic vertebral arterial stenosis, accompanied with posterior inferior cerebellum artery derived from the affected artery and related symptoms are caused/clinical benefits can be achieved through angioplasty.
* or Extracranial arterial system:
* ≥70% in the rate of stenosis with symptoms;
* nonsymptomatic patients, ≥70% in the rate of stenosis , with perfusing evidence.

Exclusion Criteria:

* >70 in age, with low rupture risk;
* stroke history in 6 weeks (contraindication for endovascular intervention);
* coexistence with intracranial tumor or AVM;
* cannot tolerant the operation;
* patient or relative refuses to participate the trail

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
morbidity rate of peri-operative cerebral hemorrhagic events | through study completion, an average of 1 year
  the morbidity rate of cerebral hemorrhagic events, with significant neuro-image evidence, during the period of treatment, including SAH/ICH/IVH caused by IAs, and intracranial hemorrhages caused by interventions focusing on AIAS
morbidity rate of peri-operative cerebral ischemic events | through study completion, an average of 1 year
  the morbidity rate of cerebral ischemic events, with significant neuro-image evidence, during the period of treatment, including all cerebral infarctions caused by interventions focusing on IAs and AIAS.

SECONDARY OUTCOMES:
Peri-operative mortality rate | through study completion, an average of 1 year
  The mortality rate during the period of treatment
Treatment-related costs | through study completion, an average of 1 year
  The total in-patient expenses of the aiming diseases, covering all treating stages
Duration of hospitalization | through study completion, an average of 1 year
  The total hospitalizations for the treatment of aiming diseases, covering all treating stages
Duration of total operating time | through study completion, an average of 1 year
  The total operating time, the sum of durations of multi-stages operation if several procedures are presented

CONTACTS AND LOCATIONS:
Overall Officials: Jizong Zhao, MD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
the IPD will be open to public researchers in 6 months after the study closed